CLINICAL TRIAL: NCT03694522
Title: FIGHT: A Phase 2 Randomized, Double-Blind, Controlled Study Evaluating Bemarituzumab (FPA144) and Modified FOLFOX6 in Patients With Previously Untreated Advanced Gastric and Gastroesophageal Junction Cancer: Phase 2 Preceded by Dose-Finding in Phase 1
Brief Title: A Study of Bemarituzumab (FPA144) Combined With Modified FOLFOX6 (mFOLFOX6) in Gastric/Gastroesophageal Junction Cancer
Acronym: FIGHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Five Prime Therapeutics, Inc. (Industry)
Collaborators: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FPA144-004 Phase 2; 2017-003507-22 (EudraCT Number); 20210113 (Other: Amgen)
Record Dates: First submitted 2018-09-14; First posted 2018-10-03 (Actual); Results first posted 2022-05-24 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — bemarituzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded (participant, treating physician)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bemarituzumab + mFOLFOX6 (Experimental): Participants received 15 mg/kg bemarituzumab administered every 2 weeks (Q2W) with a single additional bemarituzumab 7.5 mg/kg dose on cycle 1 day 8. Participants also received mFOLFOX6 chemotherapy administered Q2W. Treatment continued until unacceptable toxicity, disease progression, or death.
  Interventions: Biological: Bemarituzumab; Drug: Modified FOLFOX6
- Placebo + mFOLFOX6 (Placebo Comparator): Participants received placebo for bemarituzumab administered every 2 weeks with a single additional placebo dose on cycle 1 day 8. Participants also received mFOLFOX6 chemotherapy administered Q2W. Treatment continued until unacceptable toxicity, disease progression, or death.
  Interventions: Drug: Placebo; Drug: Modified FOLFOX6

INTERVENTIONS:
Biological: Bemarituzumab — Administered by intravenous infusion over approximately 30 minutes
  Other Names: FPA144; AMG 552
  Arms: Bemarituzumab + mFOLFOX6
Drug: Placebo — Administered by intravenous infusion over approximately 30 minutes
  Arms: Placebo + mFOLFOX6
Drug: Modified FOLFOX6 — mFOLFOX6 regimen consists of the following:
  * Oxaliplatin 85 mg/m² IV infusion over 120 minutes
  * Leucovorin 400 mg/m² IV infusion over 120 minutes, or 200 mg/m² levo-leucovorin if leucovorin is unavailable
  * 5-fluorouracil (5-FU) 400 mg/m² bolus over approximately 5 minutes then 5-FU 2400 mg/m² as a continuous IV infusion over approximately 48 hours
  Other Names: mFOLFOX6

SUMMARY:
The main objective of the Phase 2 part of the study is to evaluate the efficacy of bemarituzumab (FPA144), a targeted antibody, in combination with modified FOLFOX6 compared to placebo in combination with modified FOLFOX6 in participants with advanced gastrointestinal cancer.

DETAILED DESCRIPTION:
Study FPA144-004 is a phase 1/2, multicenter, global, double-blind, randomized, controlled study designed to evaluate the safety, tolerability, efficacy, and pharmacokinetics (PK) of bemarituzumab in combination with mFOLFOX6, compared with placebo in combination with mFOLFOX6, in adults with unresectable, locally advanced, or metastatic gastric cancer including cancer of the gastroesophageal junction (GEJ).

This study includes a Phase 1 safety run-in portion and a Phase 2 portion. The Phase 1 safety run-in is an open-label dose-escalation of bemarituzumab + mFOLFOX6 in patients with GI tumors (not FGFR2 selected) that is reported separately (NCT03343301).

The Phase 2 portion of the study (to follow the Phase 1 safety run-in) is described in this record.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically documented gastric or gastroesophageal junctional adenocarcinoma (not amenable to curative therapy)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Adequate hematological, liver and kidney function. Measurable or non-measurable, but evaluable disease using RECIST v1.1
* Fibroblast growth factor receptor 2b (FGFR2b) overexpression as determined by a centrally performed immunohistochemistry tissue test and/or FGFR2 gene amplification as determined by a centrally performed circulating tumor deoxyribonucleic acid (ctDNA) blood based assay
* Candidate for mFOLFOX6 chemotherapy

Key Exclusion Criteria:

* Untreated or symptomatic central nervous system (CNS) metastases
* Clinically significant cardiac disease,
* Peripheral sensory neuropathy >/= Common Terminology Criteria for Adverse Events (CTCAE) Grade 2
* Active infection requiring systemic treatment
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or known active or chronic hepatitis B or C infection
* Prior treatment with any selective inhibitor of the fibroblast growth factor (FGF)-FGFR pathway
* Known abnormalities of the cornea that may pose an increased risk of developing a corneal ulcer
* Known positivity for human epidermal growth factor receptor 2 (HER2)
* Women who are pregnant or breastfeeding

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2022-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (189):
- United States (29):
  - University of Arizona Cancer Center, Tucson, Arizona
  - The Oncology Institute of Tuscon, Tucson, Arizona
  - Marin Cancer Care, Inc-California Cancer Care A Medical Group, Inc, Greenbrae, California
  - Sutter Medical Group, Sacramento, California
  - UCLA Medical Centre - Santa Monica Hematology and Oncology, Santa Monica, California
  - Innovative Clinical Research Institute (ICRI), Whittier, California
  - Yale Cancer Center, New Haven, Connecticut
  - Hartford Healthcare Cancer Institute at The Hospital of Central Connecticut, Plainville, Connecticut
  - University of Chicago, Chicago, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - University of Kansas Medical Center, Westwood, Kansas
  - Oschsner Clinic Foundation, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center-Henry Ford Cancer Center, Detroit, Michigan
  - Summit Medical Group. Morristown Oncology, Morristown, New Jersey
  - University of Rochester Medical Center (URMC) - Wilmot Cancer Institute (WCI) (James P. Wilmot Cancer Center), Rochester, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - Westchester Institute For Treatment Of Cancer & Blood Disorders, White Plains, New York
  - UNC- Chapel Hill, Chapel Hill, North Carolina
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - St. Luke's Physician Group - St. Luke's Cancer Care Associates, Bethlehem, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Arlington Cancer Center, Arlington, Texas
  - Utah Cancer Specialists (Intermountain Hematology - Oncology Associates) UCS Cancer Center, South Salt Lake, Utah
  - Virginia Mason Seattle Main Clinic, Seattle, Washington
- Australia (3):
  - Chris O'brien Lifehouse, Camperdown
  - The Townsville Hospital, Douglas
  - Sydney Adventist Hospital, Wahroonga
- Belgium (4):
  - AZ Sint Jan, Bruges
  - CH de l'Ardenne, Libramont
  - CHC Clinique Saint-Joseph, Liège
  - CHU UCL Namur, site Godinne, Yvoir
- China (26):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Shiyan Taihe Hospital, Shiyan, Hubei
  - Wuhan Union Hospital of China, Wuhan, Hubei
  - The 81st Hospital of Chinese PLA, Nanjing, Jiangsu
  - Beijing Cancer Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Sino Japanese Friendship Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - Xiangya Hospital of Central South University, Changsha
  - Chongqing Daping Hospital, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Sir Run Run Shaw Hospital, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hopsital, Harbin
  - Nanton Tumor Hospital, Nantong
  - Shanghai East Hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Ruijin Hospital Affiliated to Shanghai Jiatong University School of Medicine, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou
  - Liaoning Cancer Hospital, Shenyang
  - Fourth Hospital of Hebei Medical University, Shijiazhuang
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Henan Cancer Hospital, Zhengzhou
- France (7):
  - CHRU Jean MINJOZ, Besançon
  - Chu Morvan - Institut de Cancerologie, Brest
  - Hopital Nord France Comte - Site Le Mittan, Montbéliard
  - Polyclinique de Gentilly, Nancy
  - CHU de Saint Etienne, Saint-Etienne
  - Centre de Radiotherapie - Clinique Sainte Anne, Strasbourg
  - Centre Paul Strauss, Strasbourg
- Germany (7):
  - Klinik fur Innere Medizin, Shwerpunkt Gastroenterologie, Hamatologie, Onkologie, Nephrologie, Berlin
  - Stadtisches Klinikum Braunschweig, Braunschweig
  - Krankenhaus Nordwest gGmbH, Institut fur Klinisch-Onkologische Forschung, Frankfurt am Main
  - Klinikum Ludwigsburg, Ludwigsburg
  - Universitatsmedizin Manheim, II. Medizinische Klinik, Mannheim
  - Klinikum Ostalb, Stauferklinikum Schwabisch Gmund, Zentrum fur Innere Medizin, Mutlangen
  - Kliniken Nordoberpfalz AG, Klinikum Weiden, Medizinische Klinik I, Oberpfalz
- Hungary (6):
  - National Institute of Oncology, Budapest
  - Del-Pesti Centrumkorhaz - Orszangos Hematologiai es Infektologiai Intezet, Onkologiai Osztaly, Budapest
  - Sugarterapias es Klinikai Onkologaiai Intezet B-A-Z Megyei Korhaz, Miskolc
  - Josa Andras Teaching Hospital, Nyíregyháza
  - University of Pecs, Clinic of Oncotherapy, Pécs
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz - Rendelointezet, Szolnok
- Italy (19):
  - AOU Ospedall Riuniti Umberto, Ancona
  - AO "S.G. Moscati", Avellino
  - Centro di Riferimento Oncologico, Aviano
  - Azienda Ospedaliera Spedali Civili di Brescia-Universita degli Studi Di Brescia, Brescia
  - Istituto di Ricovero e Cura a Carattere Scientifico - IRCCS di Candiolo, Candiolo
  - Azienda Socio-Sanitaria Territoriale di Cremona, Cremona
  - Azienda Ospedaliero Universitaria Caregg - I S.O.D. Oncologia Medica, Florence
  - Ospedale Policlinico S. Martino, Genova
  - Ospedale Generale Mater Salutis" - Azienda ULSS n. 21 di Legnago, Legnago
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Istituto Europeo di Oncologia, Milan
  - Servizio Oncologia Medica ed Ematologia, AOU dell'Universita, Napoli
  - Fondazione Irccs Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Policlinico Universitario Campus Bio-Medico di Roma, Roma
  - Fondazione IRCSS Casa Sollievo Della Sofferenza, San Giovanni Rotondo
  - ASST della Valtellina e dell'Alto Lario - PO di Sondrio, Sondrio
  - A.O.U. Citta della Salute e della Scienza di Torino - Presidio Molinette, Torino
  - Azienda Sanitaria Universitaria Integrata de Udine, Udine
- Japan (11):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Bunkyō City
  - Hiroshima Citizens Hospital, Hiroshima
  - St. Marianna University School of Medicine Hospital, Kawasaki
  - Japan Community Health Care Organization Kyushu Hospital, Kitakyushu
  - The Cancer Institute Hospital of JFCR, Kōtoku
  - Niigata Cancer Center Hospital, Niigata
  - Hyogo College of Medicine College Hospital, Nishinomiya
  - Osaka General Medical Center, Osaka
  - Osaka Medical College Hospital, Osaka
- Poland (8):
  - Beskidzkie Centrum Onkologii - Szpital Miejski im. Jana Pawla II w Bielsku-Bialej, Bielsko-Biala
  - Szpital Specjalistyczny w Brzozowie, Podkarpacki Osrodek Onkologiczny, Brzozów
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 w Lublinie, Lublin
  - SP ZOZ Ministerstwa Spraw Wewnetrznych z Warminsko - Mazurskim Centrum Onkologii, Olsztyn
  - Europejskie Centrum Zdrowia Otwock Szpital im. F. Chopina, Otwock
  - Lekarz Beata Madej Mruk I Partner. Spolka Partnerska Oddzial nr 1 w Rzesowie, Rzeszów
  - Wojskowy Instytut Medyczny, Centralny Szpital Kliniczny Ministerstwa Obronty Narodowej, Warsaw
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie Klinika Onkologi I Radioterapii, Warsaw
- Portugal (7):
  - Centro Hospitalar do Baixo Vouga, EPE, Aveiro
  - Hospital de Braga, Braga
  - Hospital Senhora Da Oliveira EPE, Guimarães
  - Centro Hospitalar Universitario do Porto E.P.E, Porto
  - Instituto Portugues de Oncologia do Porto Francisco Gentil E.P.E, Porto
  - Centro Hospitalar de Entre o Douro e Vouga EPE, Santa Maria da Feira
  - Unidade Local de Saude de Matosinhos EPE, Senhora da Hora
- Romania (7):
  - Institutul Clinic Fundeni - Clinica Pediatrie, Bucharest
  - Institutul Oncologic, Prof. Dr. I. Chiricuta Cluj-Napoca, Cluj-Napoca
  - S.C. Medisprof S.R.L, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta ,,Sf. Apostol Andrei" Constanta, Clinica Oncologie Medicala, Constanța
  - S.C. Centrul de Oncologie Sf. Nectarie S.R.L., Oncologie Medicala, Craiova
  - SC Oncolab SRL, Oncologie, Craiova
  - S.C. Oncocenter Oncologie Clinica S.R.L, Timișoara
- South Korea (16):
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul, Gangnam
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Kyungpook National University Chilgok Hospital, Daegu, Gyeongsangbuk-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Gachon University Gil Medical Center, Incheon, Namdong-gu
  - Dong-A University Hospital, Busan
  - Chungnam National University Hospital (CNUH), Daejeon
  - Korea University Anam Hospital, Seoul
  - Yonsei University Health System, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Spain (17):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Universitario Fundacion Alcorcon, Alcorcón
  - Hospital del Mar, Barcelona
  - Hospital Duran I Reynals - Instituto Catalan de Oncologia, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital General de Catalunya, Barcelona
  - Institut Catala d'Oncologia - Hospital Doctor Josep Trueta, Girona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Clinica Universidad de Navarra, Pamplona
  - Complejo Hospital De Navarra, Pamplona
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Hosptial Universitario Virgen Macarena, Servilla
  - Hospital Universitario Mutua de Terrassa, Terrassa
- China Medical University Hospital, Taichung, Taiwan
- Thailand (5):
  - Faculty of Medicine, Chulalongkorn University, Bangkok
  - Chiangrai Prachanukroh Hospital, Chiang Rai
  - Faculty of Medicine, Prince of Sonkla University, Hat Yai
  - Khon Kaen Hospital, Khon Kaen
  - Lampang Cancer Hospital, Lampang
- Turkey (Türkiye) (15):
  - Cukurova University Faculty of Medicine Paediatric Nephrology, Adana
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Ankara Oncology Education and Research Hospital, Ankara
  - Ondokuz Mayis University Medicine Faculty, Atakum
  - Adnan Menderes Universitesi Uygulama ve Arastirma Hastanesi, Aydin
  - Uludag Universitesi Tip Fakultesi, Bursa
  - Gaziantep Universitesi Tip Fakultesi, Sahinbey Onkoloji Hastanesi, Gaziantep
  - Bezmialem Vakif Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Istanbul Madeniyet Universitesi Tip Fakultesi, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Medical Park Izmir Hastanesi, Izmir
  - Ege University Hopsital, Izmir
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Inonu Universitesi Tip Fakultesi Turgut Ozal Tip Merkezi, Malatya
  - Yuzuncuyil Universitesi Tip Fakultesi, Van
- Ninewells Hospital and Medical School, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wainberg ZA, Kang YK, Lee KW, Qin S, Yamaguchi K, Kim IH, Saeed A, Oh SC, Li J, Turk HM, Teixeira A, Hitre E, Udrea AA, Cardellino GG, Sanchez RG, Zahlten-Kumeli A, Taylor K, Enzinger PC. Bemarituzumab as first-line treatment for locally advanced or metastatic gastric/gastroesophageal junction adenocarcinoma: final analysis of the randomized phase 2 FIGHT trial. Gastric Cancer. 2024 May;27(3):558-570. doi: 10.1007/s10120-024-01466-w. Epub 2024 Feb 3. PMID 38308771
- [Derived] Wainberg ZA, Enzinger PC, Kang YK, Qin S, Yamaguchi K, Kim IH, Saeed A, Oh SC, Li J, Turk HM, Teixeira A, Borg C, Hitre E, Udrea AA, Cardellino GG, Sanchez RG, Collins H, Mitra S, Yang Y, Catenacci DVT, Lee KW. Bemarituzumab in patients with FGFR2b-selected gastric or gastro-oesophageal junction adenocarcinoma (FIGHT): a randomised, double-blind, placebo-controlled, phase 2 study. Lancet Oncol. 2022 Nov;23(11):1430-1440. doi: 10.1016/S1470-2045(22)00603-9. Epub 2022 Oct 14. PMID 36244398
- [Derived] Xiang H, Liu L, Gao Y, Ahene A, Macal M, Hsu AW, Dreiling L, Collins H. Population pharmacokinetic analysis of phase 1 bemarituzumab data to support phase 2 gastroesophageal adenocarcinoma FIGHT trial. Cancer Chemother Pharmacol. 2020 Nov;86(5):595-606. doi: 10.1007/s00280-020-04139-4. Epub 2020 Sep 23. PMID 32965540

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study FPA144-004 was a Phase 1/2 study. Phase 1 was a safety run-in to determine the recommended dose of bemarituzumab to be administered in combination with a fixed dose of modified FOLFOX 6 (mFOLFOX6) chemotherapy regimen in the phase 2 part of the study. Phase 1 study details and results are reported separately (NCT03343301); Phase 2 study results are reported below.
Pre-assignment Details: Participants were randomized equally to one of two treatment groups stratified based on the following factors:
  * Geographic region: United States/European Union, China, or Rest of Asia
  * Prior treatment status: de novo (no prior adjuvant/neo-adjuvant therapy) or prior adjuvant/neo-adjuvant therapy
  * Administration of a single dose of mFOLFOX6 prior to enrollment: Yes or No.
Groups:
- Bemarituzumab + mFOLFOX6: Participants received 15 mg/kg bemarituzumab administered every 2 weeks (Q2W) with a single additional bemarituzumab 7.5 mg/kg dose on cycle 1 day 8. Participants also received modified FOLFOX (mFOLFOX6) chemotherapy administered Q2W. Treatment continued until unacceptable toxicity, disease progression, or death.
- Placebo + mFOLFOX6: Participants received placebo for bemarituzumab administered Q2W with a single additional placebo dose on cycle 1 day 8. Participants also received mFOLFOX6 chemotherapy administered Q2W. Treatment continued until unacceptable toxicity, disease progression, or death.
Period: Overall Study
Arm/Group | Bemarituzumab + mFOLFOX6 | Placebo + mFOLFOX6
Started | 77 | 78
Received Any Study Treatment | 76 | 77
Completed | 15 | 12
Not Completed | 62 | 66
Not completed — Withdrawal by Subject | 8 | 10
Not completed — Physician Decision | 53 | 54
Not completed — Other | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population includes all participants who were randomized in the study.
Groups:
- Bemarituzumab + mFOLFOX6: Participants received 15 mg/kg bemarituzumab administered Q2W with a single additional bemarituzumab 7.5 mg/kg dose on cycle 1 day 8. Participants also received mFOLFOX6 chemotherapy administered Q2W. Treatment continued until unacceptable toxicity, disease progression, or death.
- Total: Total of all reporting groups
Arm/Group | Bemarituzumab + mFOLFOX6 | Placebo + mFOLFOX6 | Total
Number analyzed (Participants) | 77 | 78 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 53 | 111
  >=65 years | 19 | 25 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (11.11) | 59.1 (12.04) | 58.5 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 19 | 44
  Male | 52 | 59 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 74 | 75 | 149
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 45 | 44 | 89
  Black or African American | 0 | 1 | 1
  American Indian or Alaska Native | 0 | 1 | 1
  White | 30 | 31 | 61
  Other | 2 | 1 | 3
Geographic Region [Count of Participants; unit: Participants] — European Union (EU) includes Italy, Turkey, Spain, Portugal, Hungary, Germany, France, Romania, Poland, and the United Kingdom.
  Rest of Asia includes Japan, Taiwan, and South Korea.
  Participants
    United States / European Union | 32 | 34 | 66
    China | 14 | 13 | 27
    Rest of Asia | 31 | 31 | 62
Prior Treatment Status [Count of Participants; unit: Participants]
  Prior adjuvant/neo-adjuvant therapy | 14 | 13 | 27
  No prior adjuvant/neo-adjuvant therapy | 63 | 65 | 128
Administration of a Single Dose of mFOLFOX6 Prior to Enrollment [Count of Participants; unit: Participants]
  Yes | 35 | 36 | 71
  No | 42 | 42 | 84
Site of Primary Cancer [Count of Participants; unit: Participants]
  Gastric cancer | 66 | 71 | 137
  Gastroesophageal junction cancer | 11 | 7 | 18
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale to assess a patient's disease status.
  * 0 = Fully active, able to carry out all pre-disease performance without restriction;
  * 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature;
  * 2 = Ambulatory and capable of all self-care, unable to carry out any work activities. Up and about > 50% of waking hours;
  * 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours;
  * 4 = Completely disabled, confined to bed or chair;
  * 5 = Dead.
  Participants
    0 (Fully active) | 25 | 28 | 53
    1 (Restricted activity but ambulatory) | 52 | 50 | 102

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as time from randomization until the date of radiographic disease progression based on investigator assessment using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or death from any cause, whichever came first. PFS was analyzed using Kaplan-Meier methods. Participants with no progression or death, or who started new anticancer therapy before documented progression or death without documented progression, or who had ≥ 2 consecutive missing tumor assessments before documented progression or death without documented progression were censored on the date of last adequate tumor assessment. Participants with no baseline tumor assessment, were censored at the date of randomization.
  The primary efficacy analysis was pre-specified to be conducted after at least 84 PFS events were observed.
Time Frame: From randomization until the primary analysis data cut-off date of 23 September 2020; median time on follow-up was 10.9 months.
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bemarituzumab + mFOLFOX6 | Placebo + mFOLFOX6
Number analyzed (Participants) | 77 | 78
months | 9.5 [7.3 to 12.9] | 7.4 [5.8 to 8.4]
Statistical Analysis 1: Comparison: Bemarituzumab + mFOLFOX6 vs Placebo + mFOLFOX6; Test type: Superiority; p = 0.0727, Stratified log-rank test; Adjusted for randomization stratification factors of geographic region and administration of mFOLFOX6 single dose prior to randomization; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.44 to 1.04] — Hazard ratio and 95% CIs were calculated using the Cox proportional hazards model, adjusted for randomization stratification factors, including geographic region and administration of mFOLFOX6 single dose prior to randomization

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from randomization until death from any cause. Participants who were lost to follow-up or did not have a date of death were censored at the last date that they were known to be alive. Participants with confirmed death or alive status after the data cutoff date were censored at the data cutoff date. Median OS was estimated using a Kaplan-Meier analysis.
Time Frame: as for outcome 1
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bemarituzumab + mFOLFOX6 | Placebo + mFOLFOX6
Number analyzed (Participants) | 77 | 78
months | NA [13.8 to NA] — Could not be estimated due to the low number of events | 12.9 [9.1 to 15.0]
Statistical Analysis 1: Comparison: Bemarituzumab + mFOLFOX6 vs Placebo + mFOLFOX6; Test type: Superiority; p = 0.0268, Stratified log-rank test; Adjusted for randomization stratification factors, including geographic region and administration of mFOLFOX6 single dose prior to randomization; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.35 to 0.95] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Tumor response assessment was performed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guidelines. ORR is defined as the percentage of participants who achieved a best overall response (BOR) of either complete response (CR) or partial response (PR) based on investigator assessment of tumor lesions per RECIST v1.1.
  CR was defined as the disappearance of all lesions except lymph node short axis < 10 mm; PR was defined as a ≥ 30% reduction in sum of diameters in target lesions.
Time Frame: Tumor assessments were performed every 8 weeks until 12 months and then every 12 weeks thereafter until disease progression or additional anticancer therapy was initiated; the median duration of follow-up time was 10.9 months.
Population: Intent-to-treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bemarituzumab + mFOLFOX6 | Placebo + mFOLFOX6
Number analyzed (Participants) | 77 | 78
percentage of participants | 46.8 [35.3 to 58.5] | 33.3 [23.1 to 44.9]
Statistical Analysis 1: Comparison: Bemarituzumab + mFOLFOX6 vs Placebo + mFOLFOX6; Test type: Superiority; p = 0.1060, Cochran-Mantel-Haenszel; P-value was calculated based on stratum-adjusted Cochran-Mantel-Haenszel (CMH) proportions; Difference = 13.1, 95% CI 2-sided [-2.8 to 29.0]

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs are defined as adverse events (AEs) that started or worsened from the start of study drug to 28 days after permanent discontinuation of study drug.
  A serious AE is defined as any untoward medical occurrence that:
  * Resulted in death;
  * Was life-threatening;
  * Required inpatient hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent or significant disability or incapacity;
  * Was a congenital anomaly or birth defect.
  The investigator assessed the causality/relationship between study treatment and each AE, and assessed the severity of each AE according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 5.0 on a scale from mild (Grade 1), moderate (Grade 2), severe (Grade 3), life-threatening (Grade 4), or death due to the AE (Grade 5). Cornea and retina AEs were defined by Standardized Medical Dictionary for Regulatory Activities Queries (SMQs) of corneal disorders and retinal disorders (broad).
Time Frame: From first dose of study drug to 28 days after last dose of study drug. Actual median (min, max) duration of treatment emergent period was 29 (4.1, 157) weeks in the bemarituzumab + mFOLFOX6 group and 28 (4.3, 133) weeks in the placebo + mFOLFOX6 group.
Population: Safety population includes all participants who received any portion of at least 1 dose of study treatment (bemarituzumab + mFOLFOX6 or placebo + mFOLFOX6).
Measure: Count of Participants; unit: Participants
Arm/Group | Bemarituzumab + mFOLFOX6 | Placebo + mFOLFOX6
Number analyzed (Participants) | 76 | 77
Participants
  Any treatment-emergent adverse event (TEAE) | 76 | 76
  TEAE with Grade ≥ 3 | 63 | 58
  TEAE related to any study drug | 72 | 73
  TEAE with Grade ≥ 3 related to any study drug | 57 | 48
  Serious adverse event (SAE) | 26 | 28
  SAE related to any study drug | 11 | 15
  TEAE leading to discontinuation of bemarituzumab/placebo | 31 | 4
  TEAE leading to discontinuation of any component of mFOLFOX6 | 35 | 29
  TEAE leading to dose reduction of bemarituzumab/placebo | 9 | 7
  TEAE leading to dose reduction of any agent of mFOLFOX6 | 48 | 44
  TEAE leading to dose delay of bemarituzumab/placebo | 51 | 41
  TEAE leading to dose delay of any agent of mFOLFOX6 | 54 | 44
  TEAE leading to Infusion interruption of bemarituzumab/placebo | 3 | 3
  TEAE leading to infusion interruption of any agent of mFOLFOX6 | 10 | 17
  Corneal disorders (SMQ) TEAE | 51 | 8
  Corneal disorders (SMQ) TEAE with Grade ≥ 3 | 21 | 0
  Corneal disorders (SMQ) TEAE related to bemarituzumab/placebo | 46 | 7
  Corneal disorder (SMQ) TEAE leading to discontinuation of bemarituzumab/placebo | 24 | 0
  Retinal disorders (SMQ) TEAE | 18 | 7
  Retinal disorders (SMQ) TEAE with Grade ≥ 3 | 1 | 0
  Retinal disorders (SMQ) TEAE related to bemarituzumab/placebo | 12 | 5
  Retinal disorder (SMQ) TEAE leading to discontinuation of bemarituzumab/placebo | 2 | 0
  TEAE leading to death (Grade 5) | 5 | 4

5. Post Hoc Outcome: Overall Survival - Updated Analysis
Description: OS is defined as time from randomization until death from any cause. Participants who were lost to follow-up or did not have a date of death were censored at the last date that they were known to be alive. Median OS was estimated using a Kaplan-Meier analysis.
Time Frame: From randomization until 28 February 2021; median time on follow-up was 12.5 months.
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bemarituzumab + mFOLFOX6 | Placebo + mFOLFOX6
Number analyzed (Participants) | 77 | 78
months | 19.2 [13.6 to NA] — Could not be estimated due to the low number of events at the time of the data cut. | 13.5 [9.3 to 15.9]
Statistical Analysis 1: Comparison: Bemarituzumab + mFOLFOX6 vs Placebo + mFOLFOX6; Test type: Superiority; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.38 to 0.94] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: All-cause mortality: From randomization until the end of study; median (min, max) time on study was 69.6 (0.1, 176.1) weeks in the Bemarituzumab + mFOLFOX6 group and 47.7 (0.6, 172.9) weeks in the Placebo + mFOLFOX6 group. Adverse Events: From first dose of any study drug to 28 days after last dose; actual median (min, max) duration of treatment emergent period was 29.4 (4.1, 157.0) weeks in the Bemarituzumab + mFOLFOX6 group and 28.3 (4.3, 133.0) weeks in the Placebo + mFOLFOX6 group.
Description: All-cause mortality is reported for all participants randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Bemarituzumab + mFOLFOX6 | Placebo + mFOLFOX6
All-Cause Mortality (participants affected / at risk) | 53/77 | 55/78
Serious Adverse Events (participants affected / at risk) | 26/76 | 28/77
Other Adverse Events (participants affected / at risk) | 75/76 | 75/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bemarituzumab + mFOLFOX6 (N=76) | Placebo + mFOLFOX6 (N=77)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 2 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 0 | 2
Death (General disorders) | 0 | 1
Incarcerated hernia (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 3
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Biliary tract infection (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 3
Pneumonia aspiration (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 2
Transaminases increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 2
White blood cell count increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Headache (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Device issue (Product Issues) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bemarituzumab + mFOLFOX6 (N=76) | Placebo + mFOLFOX6 (N=77)
Anaemia (Blood and lymphatic system disorders) | 25 | 28
Leukopenia (Blood and lymphatic system disorders) | 8 | 9
Neutropenia (Blood and lymphatic system disorders) | 15 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 4
Cataract (Eye disorders) | 7 | 1
Corneal disorder (Eye disorders) | 4 | 0
Corneal epithelium defect (Eye disorders) | 7 | 0
Dry eye (Eye disorders) | 21 | 5
Keratitis (Eye disorders) | 11 | 1
Limbal stem cell deficiency (Eye disorders) | 6 | 0
Punctate keratitis (Eye disorders) | 10 | 2
Ulcerative keratitis (Eye disorders) | 4 | 0
Vision blurred (Eye disorders) | 13 | 1
Abdominal distension (Gastrointestinal disorders) | 4 | 6
Abdominal pain (Gastrointestinal disorders) | 17 | 20
Abdominal pain upper (Gastrointestinal disorders) | 6 | 5
Constipation (Gastrointestinal disorders) | 23 | 24
Diarrhoea (Gastrointestinal disorders) | 31 | 23
Dyspepsia (Gastrointestinal disorders) | 7 | 9
Dysphagia (Gastrointestinal disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 37 | 41
Stomatitis (Gastrointestinal disorders) | 26 | 10
Vomiting (Gastrointestinal disorders) | 23 | 23
Asthenia (General disorders) | 20 | 16
Fatigue (General disorders) | 16 | 21
Mucosal inflammation (General disorders) | 8 | 4
Oedema peripheral (General disorders) | 4 | 4
Pyrexia (General disorders) | 10 | 12
Conjunctivitis (Infections and infestations) | 5 | 2
Onychomycosis (Infections and infestations) | 4 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 6 | 7
Alanine aminotransferase increased (Investigations) | 23 | 11
Aspartate aminotransferase increased (Investigations) | 24 | 15
Blood alkaline phosphatase increased (Investigations) | 7 | 5
Blood bilirubin increased (Investigations) | 7 | 4
Blood creatinine increased (Investigations) | 2 | 4
Neutrophil count decreased (Investigations) | 31 | 33
Platelet count decreased (Investigations) | 14 | 21
Weight decreased (Investigations) | 16 | 10
Weight increased (Investigations) | 0 | 4
White blood cell count decreased (Investigations) | 16 | 12
Decreased appetite (Metabolism and nutrition disorders) | 23 | 28
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5
Dizziness (Nervous system disorders) | 6 | 4
Dysgeusia (Nervous system disorders) | 5 | 6
Headache (Nervous system disorders) | 7 | 4
Neuropathy peripheral (Nervous system disorders) | 13 | 11
Neurotoxicity (Nervous system disorders) | 3 | 5
Paraesthesia (Nervous system disorders) | 13 | 10
Peripheral sensory neuropathy (Nervous system disorders) | 15 | 15
Insomnia (Psychiatric disorders) | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 6
Nail disorder (Skin and subcutaneous tissue disorders) | 6 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 5 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 5 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 8
Rash (Skin and subcutaneous tissue disorders) | 4 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 3
Hypertension (Vascular disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The CTA generally does not restrict an investigator's discussion of trial results after completion. Amgen has limited time to review material discussing trial results (up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control/approval of content. For multicenter studies, PI agrees not to publish results before first multi-center publication for at least 18 mo after study completion at all sites & all analyses of data resulting from Study.

DOCUMENTS (2):
  • Study Protocol (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT03694522/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT03694522/SAP_001.pdf